CLINICAL TRIAL: NCT06678997
Title: Efficacy and Safety of Polaprezinc/Zinc L-carnosine (Hepilor) in Infants With Gastroesophageal Reflux
Brief Title: Polaprezinc (Zinc L-carnosine) in Infants With Gastroesophageal Reflux
Acronym: GER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Di Nardo, Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HEPILOR PED
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Gastroesophageal Reflux (GER); Infants
Keywords: Gastroesophageal Reflux; Infants; Zinc-L carnosine/Polaprezinc
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc-L carnosine/Polaprezinc (Experimental): This group will receive Zinc-L carnosine/Polaprezinc (Hepilor Liquido) 1 hour after meals: 2.5 ml twice a day in infants weighing <5 kg or 5 ml twice a day in infants weighing >5 kg.
  Interventions: Device: Zinc-L carnosine/Polaprezinc
- Thickened formula (Active Comparator): Infants will receive thickened but not hydrolyzed formula
  Interventions: Other: Thickened formula

INTERVENTIONS:
Device: Zinc-L carnosine/Polaprezinc — This will be a randomised, single blind, controlled, multicenter study, designed to evaluate efficacy and safety of Zinc-L carnosine/Polaprezinc in infants (1-12 months of age) with symptoms suggestive of GER. This study will include a 2-week screening period, and a 8-week treatment period. After the screeing phase, eligible patients will be randomly assigned to either Zinc-L carnosine/Polaprezinc (Hepilor Liquido, Azienda Farmaceutica Italiana, Italy) twice a day or thickened formula, in a 1:1 ratio, for 8 weeks. Study visits will be conducted every 4 weeks during the treatment period.
  Other Names: Zinc-L carnosine/Polaprezinc (Hepilor Liquido)
  Arms: Zinc-L carnosine/Polaprezinc
Other: Thickened formula — This will be a randomised, single blind, controlled, multicenter study, designed to evaluate efficacy and safety of Zinc-L carnosine/Polaprezinc in infants (1-12 months of age) with symptoms suggestive of GER. This study will include a 2-week screening period, and a 8-week treatment period. After the screeing phase, eligible patients will be randomly assigned to either Zinc-L carnosine/Polaprezinc (Hepilor Liquido, Azienda Farmaceutica Italiana, Italy) twice a day or thickened formula, in a 1:1 ratio, for 8 weeks. Study visits will be conducted every 4 weeks during the treatment period.
  Arms: Thickened formula

SUMMARY:
The goal of this clinical trial is to evaluate efficacy and safety of Zinc-L carnosine/Polaprezinc in infants with GER.

Researchers will compare Zinc-L carnosine/Polaprezinc to a placebo (a look-alike substance that contains no drug) to see if Zinc-L carnosine/Polaprezinc works to treat infants with GER.

Participants will:

Take drug Zinc-L carnosine/Polaprezinc or a thickened formula every day for 8 weeks Visit the clinic once every 4 weeks for checkups and questionnaires

DETAILED DESCRIPTION:
This will be a randomised, single blind, controlled, study, designed to evaluate efficacy and safety of Zinc-L carnosine/Polaprezinc in infants (1-12 months of age) with symptoms suggestive of GER. The study will include a 2-week screening period, and a 8-week parallel arms treatment period. After the screening phase, eligible patients will be randomly assigned to either thickened formula or polaprezing twice a day, in a 1:1 ratio, for 8 weeks. Study visits will be conducted every 4 weeks during the treatment period. All the subjects will be blindly allocated by means of scratch cards to one of the two treatment groups according to a computer-generated randomisation list provided by our statistician. A validated program will be used by an independent statistician to generate a randomisation list with blocks, block size=4, pre-allocated to centres. Only study investigators will be blinderd to the randomisation codes. The codes will be kept confidential until the end of the study when the randomisation code will be broken after the database lock. All subjects will undergo a formal clinical assessment. The protocol will be approved by and indipendent etichs committee and conducted according to the Declaration of Helsinki and the principles of good clinical practice.

Eligible patients with symptoms meeting Rome IV criteria for diagnosis of Infant Regurgitation will be recruited from Sant'Andrea University Hospital and from Children Hospital SS Antonio E Biagio E C. Arrigo.

The estimated total sample size that was aimed was 48 (24 children per arm) with the power of 80% (alpha of 5%). We estimated a dropout rate of 20% and aimed to recruit 60 participants to provide at least 48 evaluable assessments.

Efficacy analysis will be performed on ITT population. A sensitivity analysis on PP population will be carried out only if 5% or more ITT subjects are excluded from PP population.

Comparison between the two groups will be performed according to ANCOVA model. For all ANCOVA models, the assumptions of normality and homogeneity of variance will be investigated. Violation of these assumptions will be overcome by performing a non-parametric test (the Wilcoxon Rank Sum test).

Statistical analysis will be performed using the computer software SPSS 25.0

ELIGIBILITY:
Inclusion Criteria:

* Patients with infant regurgitation accoding to Rome IV criteria
* Healthy infants aged 1-12 months
* I-GERQ-R score ≥ 16 at baseline

Exclusion Criteria:

* Organic disease
* Current or pregress use of pharmacological treatment for gastric acid suppression or current use of thickened formula
* Past history of preterm birth or atopy
* Absence of informed consent

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
I-GERQ-R questionnaire | From enrollment to the end of treatment at 8 weeks.
  The primary outcome will be the quantitative improvement in Infant Gastroesophageal Reflux Questionnaire Revised (I-GERQ-R) score from baseline to the end of the treatment period. The total score ranges from 0 to 42. A cut-off of ≥ 16 has been suggested to discriminate between GER and GER-disease.

SECONDARY OUTCOMES:
Acceptability | From enrollement to the end of treatment at 8 weeks.
  Secondary outcome will be the evaluation of product acceptability according to a five-point Likert scale, ranges from 1 (very poor) to 5 (very good)

IPD SHARING:
Plan to Share IPD: Undecided